CLINICAL TRIAL: NCT06660329
Title: Efficacy and Safety of Tofacitinib in Patients with Refractory Blau Syndrome: a Prospective Cohort Study
Brief Title: Efficacy and Safety of Tofacitinib in Refractory Blau Syndrome
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Hongmei Song, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K6581
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Blau Syndrome
Keywords: Blau syndrome; Janus kinase inhibitors
MeSH Terms: conditions — Blau syndrome | interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Janus kinase inhibitors (Experimental): Tofacitinib is used according to weight: 5~<7kg，2mg；7~<10kg，2.5mg；10~<15kg，3mg；15~<25kg，3.5mg；25~<40kg，4mg；≥40kg，5mg. All is twice a day.
  Interventions: Drug: Janus Kinase Inhibitor

INTERVENTIONS:
Drug: Janus Kinase Inhibitor — Tofacitinib is used according to weight: 5~<7kg，2mg；7~<10kg，2.5mg；10~<15kg，3mg；15~<25kg，3.5mg；25~<40kg，4mg；≥40kg，5mg. All is twice a day.

SUMMARY:
This is a prospective cohort study to observe the efficacy and safety of Tofacitinib in children with Blau syndrome (BS). The investigators would analyze the rate of remission or low disease activity after treatment as well as changes in inflammatory markers, patients' and physician's global assessment of disease activity to determine the efficacy and safety of Tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have pathogenic mutation(s) in NOD2 gene;
* Patients who have clinical manifestations such as granulomatous dermatitis, arthritis, uveitis, vasculitis, interstitial lung disease and so on;
* Clinical remission was not achieved after ≥12 weeks of treatment with at least one immunosuppressant or biologics.

Exclusion Criteria:

Patients will not be included if meets any of the following criteria:

* Being treated with IL-1 inhibitor, or other biological agents;
* Pregnant and lactating women;
* Serious organ function failure, expected life time less than 6 months.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
rate of remission or low disease activity | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
RCB(Response in Chinese children with Blau syndrome) 30, 50, 70 response rates | From enrollment to the end of treatment at 3, 6, 9, 12 months
Changes in inflammatory markers (including erythrocyte sedimentation rate, C reactive protein), cytokines (including IL-1β, IL-6, IL-17, IL-18, TNFα, IFN γ) and expression of type I interferon-stimulated genes over baseline | From enrollment to the end of treatment at 1,3, 6, 9, 12 months
  Changes are standardized as the ratio of the numerical difference before and after treatment to the baseline value
Proportion of recurrent uveitis | From enrollment to the end of treatment at 12 months
Incidence of new organ involvement | From enrollment to the end of treatment at 1,3, 6, 9, 12 months
Number of participants with adverse effect | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided